CLINICAL TRIAL: NCT01026831
Title: A Phase III, Randomized, Active Comparator-Controlled, Twelve-Week, Double-Masked Clinical Trial to Compare the Efficacy and Safety of Preservative-Free MK2452 (0.0015%) and Preservative-Free Timolol Maleate (0.5%) in Patients With Open-Angle Glaucoma and Ocular Hypertension
Brief Title: Preservative-Free MK2452 (Tafluprost) for Open-Angle Glaucoma/Ocular Hypertension (MK2452-001)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2452-001; 2009_701
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tafluprost (Experimental): Preservative-free tafluprost
  Interventions: Drug: Preservative-Free Tafluprost
- timolol maleate (Active Comparator): Preservative-free timolol maleate
  Interventions: Drug: Comparator: timolol

INTERVENTIONS:
Drug: Preservative-Free Tafluprost — One drop of preservative-free vehicle per eye in the morning, and one drop of preservative-free tafluprost (0.0015%) per eye in the evening for 12 weeks
  Other Names: MK2452
  Arms: Tafluprost
Drug: Comparator: timolol — One drop of preservative-free timolol maleate (0.5%) per eye twice daily for 12 weeks
  Arms: timolol maleate

SUMMARY:
This study was to compare the safety and efficacy of the preservative-free formulation of 0.0015% MK2452 (tafluprost) and preservative-free 0.5% timolol maleate in patients with open-angle glaucoma and ocular hypertension. This study was to demonstrate that the preservative-free formulation of 0.0015% tafluprost is non-inferior to preservative-free 0.5% timolol maleate.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with primary open-angle glaucoma, pigmentary glaucoma, capsular glaucoma/pseudoexfoliation, or ocular hypertension
* Patient has a mean (or median) IOP of >=23 and =<36 in at least one eye at the 0800 hours time point at the Baseline Visit.
* Patient has <5 mmHg difference in mean (or median) IOP between eyes at each time point (0800 hours, 1000 hours, and 1600 hours) at Baseline.
* Patient is currently using a prescribed ocular hypotensive medication and has been on a stable dose for 30 days prior to screening, or patient is drug-naive (those who have never used or who have not used ocular hypotensive medication for at least 4 weeks prior to screening)
* Patient is able to safely discontinue current ocular hypotensive medication during up to the 4-week washout period
* Patient has vision corrected to 20/80 or better in each eye
* Patient is willing and able to avoid wearing contact lenses from 4 weeks prior to dosing through 24 hour after final dosing
* Patient is willing and able to self-administer or has an able person available on a daily basis to assist with administration of study medications
* Patient is not pregnant and not planning to become pregnant during the study
* Patient is male or female ≥18 of age on the day of signing the informed consent

Exclusion Criteria:

* Patient is unable to use study medication in the affected eye(s)
* Patient has a history of inflammatory ocular surface disease or anterior or posterior uveitis in either eye
* Patient has a history of retinal detachment, diabetic retinopathy, or other progressive retinal disease
* Patient has experienced significant visual field loss within the last year
* Patient has had intraocular surgery in either eye in the last 4 months
* Patient has a history of glaucoma surgery or refractive surgery in either eye
* Patient is currently taking two or more anti-glaucoma medications (except Cosopt™ or its generic formulation)
* Patient has previously used tafluprost
* Patient has a history of cardiovascular disorder within 6 months prior to screening
* Patient has a history of bronchial asthma, wheezing, pneumonia, COPD, other pulmonary disease, or abnormal chest x-ray
* Patient has a mean (or median) IOP >36 mmHg in either eye at the Screening Visit or at any time point (0800 hours, 1000 hours, and 1600 hours) of the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2010-01-06 (Actual); Primary Completion 2010-09-17 (Actual); Study Completion 2010-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Chabi A, Varma R, Tsai JC, Lupinacci R, Pigeon J, Baranak C, Noble L, Lines C, Ho TW. Randomized clinical trial of the efficacy and safety of preservative-free tafluprost and timolol in patients with open-angle glaucoma or ocular hypertension. Am J Ophthalmol. 2012 Jun;153(6):1187-96. doi: 10.1016/j.ajo.2011.11.008. Epub 2012 Feb 4. PMID 22310086

RESULTS

PARTICIPANT FLOW:
Groups:
- Tafluprost: One drop of preservative-free vehicle per eye in the morning, and one drop of preservative-free tafluprost (0.0015%) per eye in the evening for 12 weeks.
- Timolol Maleate: One drop of preservative-free timolol maleate (0.5%) per eye twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Tafluprost | Timolol Maleate
Started | 320 (randomized) | 323 (randomized)
Completed | 306 | 312
Not Completed | 14 | 11
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafluprost | Timolol Maleate | Total
Number analyzed (Participants) | 320 | 323 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.7) | 63.3 (11.6) | 63.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 192 | 375
  Male | 137 | 131 | 268

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) Change From Baseline at All 9 Time Points During the Study (0800, 1000 and 1600 Hrs at Weeks 2, 6, and 12)
Description: IOP was measured using a Goldmann applanation tonometer. The primary evaluation was based on the study eye (the worse eye based on the 0800 hour IOP baseline or the right eye when both eyes had the same IOP).
  IOP change from baseline was calculated using the baseline IOP at each time point (0800 hours at baseline to 0800 hours at Week 2, 6, and 12; 1000 hours at baseline to 1000 hours at Week 2, 6, and 12; 1600 hours at baseline to 1600 hours at Week 2, 6, and 12).
  Lowering elevated IOP is a treatment goal of glaucoma.
Time Frame: Baseline, Weeks 2, 6, and 12.
Population: The Per-Protocol (PP) approach excluded all patients with important protocol violations and was performed for the efficacy endpoints. The PP population excluded patients due to important deviations from the protocol that may have substantially affected the results of the primary endpoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Tafluprost | Timolol Maleate
Number analyzed (Participants) | 299 | 313
mmHg
  Week 2 - 0800 (n=280; n=295) | -7.1 [-7.5 to -6.8] | -6.8 [-7.1 to -6.5]
  Week 2 - 1000 (n=293; n=305) | -6.8 [-7.1 to -6.5] | -6.1 [-6.4 to -5.8]
  Week 2 - 1600 (n=289; n=302) | -6.2 [-6.5 to -5.9] | -5.3 [-5.7 to -5.0]
  Week 6 - 0800 (n=294; n=308) | -7.3 [-7.6 to -6.9] | -7.4 [-7.7 to -7.1]
  Week 6 - 1000 (n=298; n=312) | -7.0 [-7.3 to -6.7] | -6.6 [-6.9 to -6.3]
  Week 6 - 1600 (n=295; n=310) | -6.3 [-6.7 to -6.0] | -5.5 [-5.9 to -5.2]
  Week 12 - 0800 (n=296; n=308) | -7.4 [-7.8 to -7.1] | -7.5 [-7.8 to -7.1]
  Week 12 - 1000 (n=298; n=312) | -7.0 [-7.4 to -6.7] | -6.6 [-7.0 to -6.3]
  Week 12 - 1600 (n=295; n=310) | -6.2 [-6.5 to -5.9] | -5.7 [-6.0 to -5.4]

2. Other Pre Specified Outcome: Baseline IOP
Description: IOP was measured using a Goldmann applanation tonometer. The primary evaluation was based on the study eye (the worse eye based on the 0800 hour IOP baseline or the right eye when both eyes had the same IOP).
Time Frame: Baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Tafluprost | Timolol Maleate
Number analyzed (Participants) | 299 | 313
mmHg
  Baseline 0800 timepoint (n=299; n=313) | 26.1 [25.8 to 26.4] | 26.0 [25.7 to 26.2]
  Baseline 1000 timepoint (n=299; n=313) | 24.8 [24.5 to 25.2] | 24.6 [24.2 to 24.9]
  Baseline 1600 timepoint (n=296; n=312) | 23.8 [23.4 to 24.2] | 23.5 [23.2 to 23.9]

ADVERSE EVENTS:
Arm/Group | Tafluprost | Timolol Maleate
Serious Adverse Events (participants affected / at risk) | 2/320 | 7/323
Other Adverse Events (participants affected / at risk) | 0/320 | 0/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafluprost (N=320) | Timolol Maleate (N=323)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
retinal detachment (Eye disorders) | 0 (0) | 1 (1)
colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
hernia (General disorders) | 0 (0) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.